CLINICAL TRIAL: NCT04871503
Title: Simultaneous Application of High-Intensity Focused Electromagnetic Procedure and Radiofrequency for Toning of Buttocks
Brief Title: High-Intensity Focused Electromagnetic Procedure and Radiofrequency for Toning of Buttocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899_300
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Muscle Tone

STUDY DESIGN:
Intervention Model Description: The subjects will be enrolled and assigned into two study groups; HIFEM+RF (HR) and HIFEM (H) group. Subjects of both groups will be required to complete four (4) treatment visits and two follow-up visits. All of the study subjects will receive the treatment with the subject device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HIFEM+RF (HR) (Experimental): The HR group will receive treatment with intensities of a magnetic field and radiofrequency energy just below the patient's tolerance threshold. The device will induce visible muscle contractions along with mild heating of the muscles.
  Interventions: Device: BTL-899 Buttocks
- HIFEM (H) (Experimental): The H group will receive a treatment with the intensities of the magnetic field just below the patient's tolerance threshold without the use of radiofrequency.
  Interventions: Device: BTL-899 Buttocks

INTERVENTIONS:
Device: BTL-899 Buttocks — The treatment administration phase in both study groups will consist of four (4) treatments, delivered 5-10 days apart. The applicators of BTL-899 will be applied over the gluteal area.

SUMMARY:
This study will evaluate the clinical efficacy and safety of the BTL-899 device for toning of buttocks. The study is a prospective multi-center open-label two-arm study. The subjects will be enrolled and assigned into two study groups. The subjects will be enrolled and assigned into two study groups; HIFEM+RF (HR) and HIFEM (H) group. Subjects of both groups will be required to complete four (4) treatment visits and two follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Voluntarily signed an informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain her regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing, and menstruation
* Intrauterine device (IUD)
* Swollen or neoplastic tissues, space-occupying lesions or skin eruptions in the treatment area
* Basedow's disease

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
The evaluation of change in structure of subcutaneous tissues between pre-treatment and post-treatment based on MRI imaging in both study groups. | 4 months
  The evaluation of structural changes of subcutaneous tissues between pre-treatment and post-treatment based on MRI imaging through measurements of the thickness of subcutaneous tissues
The evaluation of change in adipose and muscle layer thickness. | 4 months
  The evaluation of change in adipose and muscle layer thickness between pre-treatment and post-treatment based on hip circumference measurements.

SECONDARY OUTCOMES:
Patient's satisfaction with study treatment measured via questionnaires | 4 months
  To determine the patient's satisfaction with study treatment. The 5-point Likert scale Satisfaction questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome. Subject satisfaction will be assessed after the last therapy visit and during the follow-up visits with 4therapy-related questions, where the answer "Strongly agree" will be the best possible answer and "Strongly disagree" the worst.
Evaluation of the Therapy's Safety Measured Via Therapy Comfort Questionnaire | 4 months
  On Numerical Analog Scale (0-10), where 0 represents 'no pain' and 10 represents 'worst possible pain' select the level of pain experienced during the treatment. The outcome will further be measured through the occurrence of adverse events or lack thereof.

CONTACTS AND LOCATIONS:
Overall Officials: Georgi Petkov, Study Director — Sponsor GmbH
Locations (5):
- United States (5):
  - Contour Medical, Gilbert, Arizona
  - Skin Laser and Surgery Specialist, a Division of Schweiger Dermatology, Hackensack, New Jersey
  - New Jersey Plastic Surgery (NJPS), Montclair, New Jersey
  - JUVA Skin & Laser Center, New York, New York
  - Refresh Dermatology, Houston, Texas

IPD SHARING:
Plan to Share IPD: No